CLINICAL TRIAL: NCT00980148
Title: Randomized Clinical Trial Evaluating Treatment Failure Following Recommended Therapy (Azithromycin Versus Doxycycline) for Genital Chlamydial Infection in Males and Females in Youth Correctional Facilities
Brief Title: Treatment Failure of Chlamydial Infection in Males and Females in Youth Correctional Facilities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0012
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2014-06

CONDITIONS: Chlamydial Infection
Keywords: Chlamydia trachomatis, Chlamydia, Doxycycline, Azithromycin
MeSH Terms: conditions — Chlamydia Infections | interventions — Azithromycin; Doxycycline

ARMS (2):
- Arm2 (Experimental): Doxycycline 100 mg oral twice a day (BID) for 7 days; 153 subjects
  Interventions: Drug: Doxycycline
- Arm 1 (Experimental): Azithromycin 1 gm oral single dose; 153 subjects
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — FDA approved, a 1 gm single dose, two 500 mg tablets.
  Arms: Arm 1
Drug: Doxycycline — FDA approved, a 100 mg capsule twice a day for 7 days.
  Arms: Arm2

SUMMARY:
Chlamydia is a common infection among youth and can be given from one person to another during sex. Many people who have chlamydia have no signs of infection at all, but can pass the infection to anyone they have sex with. If not treated, chlamydia can lead to serious health problems. This study will look at how well medicines given for chlamydia infection work. The study requires 306 evaluable subjects, chlamydia-positive, males and non-pregnant females, ages 12-21, living in long-term, gender-segregated youth correctional facilities. Participants will be assigned to receive either doxycycline (2 times per day, by mouth, for 7 days) or azithromycin (1 single dose by mouth). Study procedures will include collection of at least 3 urine samples to test for chlamydia. Study visits will occur during initial enrollment in the study, day 28 after starting treatment, and day 67. Participants will be involved in study related procedures for up to 67 days.

DETAILED DESCRIPTION:
Genital chlamydia is a public health concern. The World Health Organization (WHO) estimates that 90 million of all new cases of sexually transmitted diseases (STDs) per year are caused by Chlamydia (C.) trachomatis. In the United States alone, approximately 3 million new cases of chlamydia are reported yearly, and the costs associated with their management and complications exceed $2 billion. Unfortunately, at least 75 percent of females with chlamydia are asymptomatic, and unless the infection is detected through chlamydia testing (screening), their infection may be transmitted to others or lead to complications. The Centers of Disease Control and Prevention (CDC) recommends either azithromycin 1 gram (gm) by mouth (PO) once or doxycycline 100 milligrams (mg) PO twice daily (BID) for 7 days as co-equal therapies for uncomplicated chlamydia. A secondary aim will be to determine demographic predictors of chlamydia treatment failure following azithromycin or doxycycline treatment, and to explore clinical parameters, which distinguish those with persistent infection. The study design of this Phase III trial will address major limitations of prior chlamydia efficacy studies and the findings will reveal both the true efficacy of azithromycin and doxycycline in uncomplicated chlamydia in adolescents and the factors that predict treatment failure. This study is designed primarily to determine the frequency of chlamydia treatment failure following either azithromycin or doxycycline regimens and to evaluate whether the efficacy of the azithromycin regimen is inferior to the doxycycline regimen. Both drugs are Food and Drug Administration (FDA) approved for use in the U.S. The study will enroll 650 males and females age 12-21 years in good health (based on vital signs and provider's clinical evaluation documented in medical records) who are residing in long-term gender-segregated (not co-ed) youth correctional facilities (YCFs) (usual stay >3 weeks) and who are identified as chlamydia-infected would comprise the study population until 306 evaluable subjects are obtained . Only individuals who have a positive chlamydia screening test are enrolled, and those with negative screening tests are excluded. Consenting chlamydia-positive subjects at the enrollment visit (study visit 1) will be enrolled, asked to provide demographic data, to provide a first-void urine sample (not a mid-stream specimen) for repeat chlamydia testing with Gen-Probe (GP) AC2 (for verification of chlamydia), and then randomized to 1 of 2 treatment arms (190 153 subjects per arm): doxycycline 100 mg PO BID for 7 days or azithromycin 1 gm PO single dose. Both therapies are given as directly observed, and side effects are evaluated at the first follow-up visit (day 28 after study drug initiation). If a subject who's GP AC2 from the enrollment treatment visit returns negative for C. trachomatis, they will be categorized as unevaluable and will be removed from the study, then the site investigator will determine whether the subject will complete this treatment or will receive other therapy. Subjects whose GP AC2 at the enrollment treatment visit is positive for C. trachomatis will then be asked to provide a first-void urine sample for repeat chlamydia testing with GP AC2 at 28- and 67-days after study drug initiation [corresponding to the first follow-up visit (study visit 2) and second follow-up visit (study visit 3), respectively].

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 12 and 21 years
* Residing in a long-term gender-segregated (no co-ed) youth correctional facility (YCF)
* Diagnosed with genital chlamydia as determined by a screening C. trachomatis nucleic acid amplification test (NAAT)
* Anticipated length of stay at the YCF at the time of enrollment is > 3 weeks
* Willingness to provide written consent
* Willingness to comply with study procedures

Exclusion Criteria:

* Diagnosed with gonorrhea as determined by a screening Neisseria gonorrhoeae nucleic acid amplification test (NAAT)
* Clinical diagnosis of pelvic inflammatory disease (PID) or epididymitis based on review of medical records
* Known allergy to tetracyclines or macrolides
* Currently pregnant or breastfeeding
* History of photosensitivity related to doxycycline use
* Having received antimicrobial therapy with activity against C. trachomatis within 21 days of the positive chlamydia screening NAAT or in the interval between the positive screening NAAT and study enrollment
* Any concomitant infection, which requires antimicrobial therapy with activity against C. trachomatis
* Previously enrolled in this study
* Unable to swallow pills
* Other exclusion criteria, per clinician judgment, that prohibits subject from enrolling in study
* Of note, current use of oral contraceptive agents (OCPs) is not an exclusion criterion

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 567 (Actual)
Dates: Start 2009-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama Hospital - Infectious Diseases, Birmingham, Alabama
  - Los Angeles County Department of Public Health - Sexually Transmitted Disease Program, Los Angeles, California

REFERENCES:
- [Derived] Geisler WM, Uniyal A, Lee JY, Lensing SY, Johnson S, Perry RC, Kadrnka CM, Kerndt PR. Azithromycin versus Doxycycline for Urogenital Chlamydia trachomatis Infection. N Engl J Med. 2015 Dec 24;373(26):2512-21. doi: 10.1056/NEJMoa1502599. PMID 26699167

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin Arm: Azithromycin 1 gm oral single dose
- Doxycycline Arm: Doxycycline 100 mg oral twice a day for 7 days
Period: Overall Study
Arm/Group | Azithromycin Arm | Doxycycline Arm
Started | 284 | 283
Completed | 155 (Completed primary evaluation at study visit # 2 (day 28 after therapy started)) | 155 (Completed primary evaluation at study visit # 2 (day 28 after therapy started))
Not Completed | 129 | 128
Not completed — Discharged from facility | 89 | 96
Not completed — Received other antichlamydia treatment | 20 | 14
Not completed — Negative for chlamydia at enrollment | 12 | 9
Not completed — Various other reasons | 8 | 9

BASELINE CHARACTERISTICS:
Population: The per protocol population is comprised of participants who completed therapy and whose failure status could be established at the day 28 visit. Participants were considered to have completed therapy if they took a single dose of azithromycin or at least 10 of the 14 doses of doxycycline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin Arm | Doxycycline Arm | Total
Number analyzed (Participants) | 155 | 155 | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 155 | 154 | 309
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.0 (0.9) | 16.8 (1.1) | 16.9 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 56 | 109
  Male | 102 | 99 | 201
Region of Enrollment [Number; unit: participants]
  United States | 155 | 155 | 310

OUTCOME MEASURES:

1. Primary Outcome: Assess Microbiological Failure of Recommended Azithromycin and Doxycycline Regimens in Uncomplicated Chlamydia Trachomatis Infection in a Setting Where Repeat Exposure to Chlamydia-infected Persons Can be Minimized.
Description: The proportion of participants with testing by Gen-Probe Aptima Combo 2 that is positive for C. trachomatis and C. trachomatis OmpA (Major Outer Membrane Protein) genotyping reveals the baseline chlamydial strain and the repeat positive chlamydial strain to be the same genotype (i.e., concordant).
Time Frame: Study visit # 2 (Day 28 after therapy started)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Azithromycin Arm | Doxycycline Arm
Number analyzed (Participants) | 155 | 155
percentage of participants | 3.2 | 0.0
Statistical Analysis 1: Comparison: Azithromycin Arm vs Doxycycline Arm; This noninferiority study tested the null hypothesis that the failure rate of azithromycin is 5% higher than that of doxycycline against the alternative hypothesis that there is no difference between the two treatments. The one-sided 90% exact confidence interval was used to estimate the difference between the two failures rates; Test type: Non-Inferiority or Equivalence — This noninferiority study tested the null hypothesis that the failure rate of azithromycin is 5% higher than that of doxycycline against the alternative hypothesis that there is no difference between the two treatments. The treatment failure rate was assumed to be 3% for both treatments. To test this hypothesis at the one-sided 0.10 significance level with power of 0.90 required 153 study subjects per arm in the per-protocol population; Risk Difference (RD) = 3.2, 90% CI 1-sided [upper limit 5.9] — The risk difference is the percentage in the azithromycin arm with treatment failure minus the percentage in the doxycycline arm with treatment failure. Noninferiority of azithromycin would be supported if the upper 90% confidence limit is below 5%

2. Secondary Outcome: Demographical Characteristics and Clinical Parameters to Predict Treatment Outcome.
Time Frame: Baseline and study visit #2 (Day 28 after therapy is started)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) that occur after study drug administration (Study Visit 1) and through the first follow-up visit (Study Visit 2, Day 28) were recorded. AEs were followed until resolution even if this extended beyond the study-reporting period.
Description: Resolution of an AE is defined as the return to pretreatment status or stabilization of the condition with the expectation that it will remain chronic. In Sept 2010, the protocol was amended to streamline reportable AE's by limiting to GI related symptoms, vaginal irritation or itching, and dermatologic reactions.
Arm/Group | Azithromycin Arm | Doxycycline Arm
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/155
Other Adverse Events (participants affected / at risk) | 11/155 | 18/155
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin Arm (N=155) | Doxycycline Arm (N=155)
Abdominal Pain (Gastrointestinal disorders) | 6 (7) | 10 (10)
Vomiting (Gastrointestinal disorders) | 6 (6) | 10 (11)

LIMITATIONS AND CAVEATS:
The analysis of the secondary endpoint Demographical Characteristics and Clinical Parameters to Predict Treatment Outcome was limited by the small number of events and is not presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No